CLINICAL TRIAL: NCT02857556
Title: Potential Biomarkers of the Severity of Endothelial Damage in End-stage Chronic Kidney Failure Evaluated at the Initiation of Intermittent or Peritoneal Dialysis
Brief Title: Potential Biomarkers of the Severity of Endothelial Damage in End-stage Chronic Kidney Failure
Acronym: DIALYSOX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of inclusions
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GAMBERT Fd. Transpl 2013
Record Dates: First submitted 2016-08-02; First posted 2016-08-05 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: End-stage Chronic Kidney Failure
MeSH Terms: interventions — Blood Specimen Collection

ARMS (2):
- group with stage 3 kidney failure (diabetic or not) (Other)
  Interventions: Biological: Blood sample; Other: Retinal photography:
- group with stage 5 kidney failure (diabetic or not) (Other)
  Interventions: Biological: Blood sample; Other: dialyse

INTERVENTIONS:
Biological: Blood sample
Other: Retinal photography:
  Arms: group with stage 3 kidney failure (diabetic or not)
Other: dialyse
  Arms: group with stage 5 kidney failure (diabetic or not)

SUMMARY:
The principal objective of this study is to qualify markers of oxidative stress in inflammatory cells (monocytes) in patients with stage 3 kidney failure (diabetic or not), and patients with end-stage kidney failure (diabetic or not), who require dialysis. The evaluation of these markers will be done by the activation and localization of proteins implicated in vascular tone and oxidative stress in monocytes, correlated with the distribution of cholesterol sphingomyelin within planar rafts and caveolae. The aim is to describe their evolution under treatment, which could lead to interventional studies.

ELIGIBILITY:
Inclusion Criteria:

* Patient who have been informed about the research
* Patients with national health insurance cover
* Patients aged between 18 and 75 years
* Patients with stage 3 kidney failure (30 ml/min < cl creat < 59 ml/min) diabetic or not
* Patients with stage 5 kidney failure (cl creat < 15 ml/mn) diabetic or not and requiring dialysis.

Exclusion Criteria:

* Patients under guardianship
* Pregnant or breast-feeding women
* Infection (including peritonitis in peritoneal dialysis, infection of the catheter insertion site),
* Neoplastic disease,
* Systemic diseases in flare,
* Patients positive for Human Immunodeficience Virus (HIV),
* Patients on immunosuppressants
* Patients taking antioxidants (selenium, vitamin C and/or E)
* Patient on statins

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-04-17 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Activation of 5 proteins relocated in the membrane of monocytes (eNOS, iNOS, gp91phox and receptors of angiotensin II (AT1 and AT2)) within dynamic lipid structures, rafts, measured by western blot-dot blot. | at the beginning of the period Day 0, at 1 month and at 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France